CLINICAL TRIAL: NCT03429933
Title: A Double-Blind, Placebo-Controlled, Randomized, Single and Multiple Ascending Dose Study (Including Food Effect, pH Effect, and Japanese Bridging Study) of the Safety, Pharmacokinetics, and Exploratory Pharmacodynamics of Oral BMS-986278 Administration in Healthy Participants
Brief Title: A Study of Experimental Medication BMS-986278 Given to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM027-009; 2017-004136-10 (EudraCT Number)
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single Ascending Dose (Experimental): BMS-986278 or placebo
  Interventions: Drug: BMS-986278; Other: Placebo
- Multiple Ascending Dose (Experimental): BMS-986278 or placebo
  Interventions: Drug: BMS-986278; Other: Placebo

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days
Other: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to investigate experimental medication BMS-986278 given to healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants must be in good general health in the opinion of the investigator
* Body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive, at screening; BMI = weight (kg)/height (m)2
* Body weight between 55 and 105 kg, inclusive, at screening
* Female participants must have documented proof that they are not of childbearing potential
* Participants in the Japanese cohorts must be first-generation Japanese (born in Japan, not living outside of Japan for more than 10 years, and both parents are ethnically Japanese)

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding
* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or that may compromise the objectives of the study, including active, or history of, liver disease, or intestinal disorder including irritable bowel syndrome
* History or presence of malignancy including hematological malignancies; participants with a history of basal cell or squamous cell carcinoma that has been treated with no evidence of recurrence within 5 years will be allowed for inclusion, as judged by the investigator
* Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug
* Any major surgery within 6 weeks of study drug administration

Other protocol defined inclusion/exclusion criteria could apply

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing adverse events (AE), serious adverse events (SAE), death, or an AE leading to study discontinuation | Up to 30 days
Number of participants with potentially clinically significant changes in ECG parameters, vital signs, clinical laboratory parameters, or physical examinations | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution, Groningen, Netherlands
- Local Institution, London, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm